CLINICAL TRIAL: NCT02294760
Title: Long-term Efficacy of Sacral Nerve Stimulation for Irritable Bowel Syndrome. A Randomised Controlled Crossover Study
Brief Title: Long-term Sacral Nerve Stimulation for Irritable Bowel Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 44418
Record Dates: First submitted 2014-11-10; First posted 2014-11-19 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Sacral Nerve Stimulation; Symptoms; Quality of Life
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Subsensory, OFF, subsensory (Active Comparator): The stimulator is set subsensory for the first 4 weeks (90% of sensory threshold), then turned OFF for the next 4 weeks and finally set subsensory for the last 4 weeks.
  Interventions: Device: Subsensory; Device: OFF
- Subsensory, subsensory, OFF (Active Comparator): The stimulator is set subsensory for the first 4 weeks (90% of sensory threshold), then set subsensory for another 4 weeks and finally turned OFF for the last 4 weeks.
  Interventions: Device: Subsensory; Device: OFF

INTERVENTIONS:
Device: Subsensory — The stimulation is set to 90% of the sensory threshold.
  Other Names: Device: External pacemaker, model 3625, Medtronic Inc.
Device: OFF — The stimulation is turned OFF.
  Other Names: Device: External pacemaker, model 3625, Medtronic Inc.

SUMMARY:
A recent randomised, controlled, crossover study has shown that sacral nerve stimulation (SNS) significantly reduces symptoms and improves quality of life of highly selected patients with irritable bowel syndrome (IBS). Relief of IBS symptoms during SNS is associated with consistent changes in rectal sensitivity and biomechanical wall properties.

The aim of the present study is to evaluate long-term efficacy of sacral nerve stimulation on symptoms and quality of life in patients with IBS in a randomised, placebo-controlled, crossover study.

DETAILED DESCRIPTION:
Twenty two patients with IBS-D or IBS-M according to the ROME III criteria, will be enrolled by invitation in the study.

Having meet inclusion criteria, the patients are first set subsensory for 4 weeks and then randomised to receive either OFF-subsensory or subsensory-OFF stimulation in a 4+4-week period.

During the PNE test the effect of the stimulation is evaluated by specific IBS symptom and quality of life questionnaires (GSRS-IBS and IBS-IS) and bowel habit diaries.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are psychologically stable and suitable for intervention and able to provide informed consent
* Patients who are diagnosed with IBS according to the Rome III criteria and characterised with IBS-D or IBS-M.
* Patients who have been treated with sacral nerve stimulation for a minimum of 3 years.

Exclusion Criteria:

* Other bowel diseases including inflammatory bowel disease
* Pregnant or breast feeding
* Patients who are considered unable to follow the planned programme of the study, including mentally illness or physiological instability
* Patients who are on medication with known influence on gastrointestinal motility including those for thyroid disease, diabetes mellitus, celiac disease and neurological diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The Gastrointestinal Symptom Rating Scale - Irritable Bowel Syndrome version | Change in the IBS-specific symptom score between the subsensory and the OFF period in the crossover study
  The questionnaire is filled in every week of the 12 week study period

SECONDARY OUTCOMES:
Irritable Bowel Syndrome - Impact Scale questionnaire | Change in the IBS-specific quality of life score between the subsensory and the OFF period in the crossover study
  The questionnaire is filled in every week of the 12 week study period

CONTACTS AND LOCATIONS:
Overall Officials: Janne Fassov, PhD, Principal Investigator — Surgical Research Unit, Department of Surgery P, Aarhus University Hospital
Locations (1):
- Surgical Research Unit, Department of Surgery P, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided